CLINICAL TRIAL: NCT01163617
Title: A Multicenter, Randomized, Open-Label Study of the Injection Time and Usability of the Physiolis Syringe and Autoinjector in Injection-Experienced Rheumatoid Arthritis Patients
Brief Title: The Usability and Injection Time of the Physiolis Syringe and Autoinjector in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: M12-088
Record Dates: First submitted 2010-05-04; First posted 2010-07-16 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Current/Physiolis Syringe (Experimental): Self-injection using current syringe at Week 0 (Visit 1), self-injection using Physiolis syringe at Week 2 (Visit 2) (Phase A)
  Interventions: Device: Adalimumab delivered in current syringe; Device: Adalimumab delivered in Physiolis syringe
- Physiolis/Current Syringe (Experimental): Self-injection using Physiolis syringe at Week 0 (Visit 1), self-injection using current syringe at Week 2 (Visit 2) (Phase A)
  Interventions: Device: Adalimumab delivered in current syringe; Device: Adalimumab delivered in Physiolis syringe
- Current/Physiolis Autoinjector (Experimental): Self-injection using current autoinjector at Week 0 (Visit 1), self-injection using Physiolis autoinjector at Week 2 (Visit 2) (Phase A)
  Interventions: Device: Adalimumab delivered in current autoinjector; Device: Adalimumab delivered in Physiolis autoinjector
- Physiolis/Current Autoinjector (Experimental): Self-injection using Physiolis autoinjector at Week 0 (Visit 1), self-injection using current autoinjector at Week 2 (Visit 2) (Phase A)
  Interventions: Device: Adalimumab delivered in current autoinjector; Device: Adalimumab delivered in Physiolis autoinjector
- Physiolis Autoinjector at 2° to 8°C (Experimental): Injection performed by health care provider at Week 4 (Visit 3) using Physiolis autoinjector at storage temperature (2° to 8°C) (Phase B)
  Interventions: Device: Adalimumab delivered in Physiolis autoinjector
- Current Autoinjector 2° to 8°C (Experimental): Injection performed by health care provider at Week 4 (Visit 3) using current autoinjector at storage temperature (2° to 8°C) (Phase B)
  Interventions: Device: Adalimumab delivered in current autoinjector
- Physiolis Autoinjector 20° to 27°C (Experimental): Injection performed by health care provider at Week 4 (Visit 3) using Physiolis autoinjector at room temperature (20° to 27°C) (Phase B)
  Interventions: Device: Adalimumab delivered in Physiolis autoinjector
- Current Autoinjector 20° to 27°C (Experimental): Injection performed by health care provider at Week 4 (Visit 3) using current autoinjector at room temperature (20° to 27°C) (Phase B)
  Interventions: Device: Adalimumab delivered in current autoinjector

INTERVENTIONS:
Device: Adalimumab delivered in current syringe — Pre-filled currently approved glass syringe containing 40 mg/0.8 mL adalimumab to be injected subcutaneously
  Other Names: ABT-D2E7; Humira
  Arms: Current/Physiolis Syringe; Physiolis/Current Syringe
Device: Adalimumab delivered in Physiolis syringe — Pre-filled Physiolis glass syringe containing 40 mg/0.8 mL adalimumab to be injected subcutaneously
  Other Names: ABT-D2E7; Humira
  Arms: Current/Physiolis Syringe; Physiolis/Current Syringe
Device: Adalimumab delivered in current autoinjector — Pre-filled currently approved autoinjector containing 40 mg/0.8mL adalimumab to be injected subcutaneously
  Other Names: ABT-D2E7; Humira
  Arms: Current Autoinjector 20° to 27°C; Current Autoinjector 2° to 8°C; Current/Physiolis Autoinjector; Physiolis/Current Autoinjector
Device: Adalimumab delivered in Physiolis autoinjector — Pre-filled Physiolis autoinjector containing 40 mg/0.8 mL adalimumab to be injected subcutaneously
  Other Names: ABT-D2E7; Humira
  Arms: Current/Physiolis Autoinjector; Physiolis Autoinjector 20° to 27°C; Physiolis Autoinjector at 2° to 8°C; Physiolis/Current Autoinjector

SUMMARY:
This was an open-label, Phase 2 study designed to obtain user experience data (Phase A) and injection time data (Phase B) in experienced adalimumab patients injected with the Physiolis pre-filled syringe and autoinjector used to administer adalimumab.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study consisting of 2 study phases with a total of 3 study visits, each visit occurring 2 weeks apart from each other. Phase A (User Experience) was a randomized, 2-period, cross-over phase in which single subcutaneous (SC) dose injections were administered using either the Physiolis autoinjector and current autoinjector or the Physiolis syringe and current syringe in a 1:1 ratio. Phase B (Injection Time) was a randomized, single-visit, parallel-arm phase, with injection into a test tube, and one SC injection given to participants using the Physiolis autoinjector or current autoinjector administered at 2 different temperature ranges (2° to 8°C [storage temperature] and 20° to 27°C [room temperature]). If a participant only completed Visit 1 and Visit 2, then the participant was to be replaced for Visit 3. If the participant only completed Visit 1, the participant was to be replaced for all study visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject was judged to be in good health as determined by the investigator based upon the results of medical history, laboratory profile, physical examination, chest x-ray, and a 12-lead electrocardiogram performed during Screening.
* Subject had a negative purified protein derivative (PPD) test (or equivalent) and chest x-ray (posterior-anterior and lateral view) at Screening.
* Subject has a diagnosis of moderate to severe rheumatoid arthritis and is treated with adalimumab in accordance with the FDA-approved Humira prescribing information.
* Subject must have self-administered adalimumab subcutaneous (SC) 40 mg injections every other week (eow) without interruption for at least 3 months prior to Screening.
* For the Phase A portion of the study, the subject must be able and willing to self administer SC injections in the thigh or abdomen (administration by another person was not permissible).

Exclusion Criteria:

* Subject has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives (whichever is longer) of the drug prior to the Visit 1, with the exception of adalimumab.
* Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the Visit 1 or oral anti-infectives within 14 days prior to Visit 1.
* Prior exposure to natalizumab (Tysabri®) or efalizumab (Raptiva®).
* Known hypersensitivity to adalimumab or its excipients.
* Regular use of any SC medications, with the exception of adalimumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Payne, PhD, Study Director — AbbVie
Locations (10):
- United States (10):
  - Site Reference ID/Investigator# 27144, Victorville, California
  - Site Reference ID/Investigator# 27153, Tampa, Florida
  - Site Reference ID/Investigator# 27150, Passaic, New Jersey
  - Site Reference ID/Investigator# 27143, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 27145, Wyomissing, Pennsylvania
  - Site Reference ID/Investigator# 27142, Charleston, South Carolina
  - Site Reference ID/Investigator# 27151, Jackson, Tennessee
  - Site Reference ID/Investigator# 27152, Dallas, Texas
  - Site Reference ID/Investigator# 27147, Houston, Texas
  - Site Reference ID/Investigator# 27155, Tyler, Texas

REFERENCES:
- [Background] Li Z, Easton R. Practical considerations in clinical strategy to support the development of injectable drug-device combination products for biologics. MAbs. 2018 Jan;10(1):18-33. doi: 10.1080/19420862.2017.1392424. Epub 2017 Nov 7. PMID 29035675
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew after Phase A and was replaced with a new participant prior to Phase B. Participants were re-randomized for Phase B.
Groups:
- Current Syringe First, Then Physiolis Syringe: Self-injection using current syringe at Week 0 (Visit 1), self-injection using Physiolis syringe at Week 2 (Visit 2) (Phase A)
- Physiolis Syringe First, Then Current Syringe: Self-injection using Physiolis syringe at Week 0 (Visit 1), self-injection using current syringe at Week 2 (Visit 2) (Phase A)
- Current Autoinjector First, Then Physiolis Autoinjector: Self-injection using current autoinjector at Week 0 (Visit 1), self-injection using Physiolis autoinjector at Week 2 (Visit 2) (Phase A)
- Physiolis Autoinjector First, Then Current Autoinjector: Self-injection using Physiolis autoinjector at Week 0 (Visit 1), self-injection using current autoinjector at Week 2 (Visit 2) (Phase A)
Period: Phase A (User Experience), Weeks 0 and 2
Arm/Group | Current Syringe First, Then Physiolis Syringe | Physiolis Syringe First, Then Current Syringe | Current Autoinjector First, Then Physiolis Autoinjector | Physiolis Autoinjector First, Then Current Autoinjector | Physiolis Autoinjector at 2° to 8°C | Current Autoinjector 2° to 8°C | Physiolis Autoinjector 20° to 27°C | Current Autoinjector 20° to 27°C
Started | 19 | 23 | 21 | 21 | 0 | 0 | 0 | 0
Completed | 19 | 21 | 20 | 21 | 0 | 0 | 0 | 0
Not Completed | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failed to meet inclusion criteria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Didn't meet inclusion/exclusion criteria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase B (Injection Time), Week 4
Arm/Group | Current Syringe First, Then Physiolis Syringe | Physiolis Syringe First, Then Current Syringe | Current Autoinjector First, Then Physiolis Autoinjector | Physiolis Autoinjector First, Then Current Autoinjector | Physiolis Autoinjector at 2° to 8°C | Current Autoinjector 2° to 8°C | Physiolis Autoinjector 20° to 27°C | Current Autoinjector 20° to 27°C
Started | 0 | 0 | 0 | 0 | 18 | 27 | 16 | 20
Completed | 0 | 0 | 0 | 0 | 18 | 27 | 16 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes participants from Phases A and B of the study
Arm/Group | All Study Participants
Number analyzed (Participants) | 85
Age, Customized [Number; unit: participants]
  <65 years | 62
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Participants' Overall Satisfaction With the Drug Administration Experience Using the Physiolis Syringe/Autoinjector in Comparison to the Current Syringe/Autoinjector
Description: Participant's overall satisfaction of the injection was collected on a 10-cm visual analog scale (VAS) completed by participants immediately after self-injection. 0 = extremely unsatisfied, 10 = extremely satisfied.
Time Frame: Phase A (Week 0 and Week 2)
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Current/Physiolis Syringe: Self-injection using current syringe at Week 0 (Visit 1), self-injection using Physiolis syringe at Week 2 (Visit 2)
- Physiolis/Current Syringe: Self-injection using Physiolis syringe at Week 0 (Visit 1), self-injection using current syringe at Week 2 (Visit 2)
- Current/Physiolis Autoinjector: Self-injection using current autoinjector at Week 0 (Visit 1), self-injection using Physiolis autoinjector at Week 2 (Visit 2)
- Physiolis/Current Autoinjector: Self-injection using Physiolis autoinjector at Week 0 (Visit 1), self-injection using current autoinjector at Week 2 (Visit 2)
Arm/Group | Current/Physiolis Syringe | Physiolis/Current Syringe | Current/Physiolis Autoinjector | Physiolis/Current Autoinjector
Number analyzed (Participants) | 19 | 23 | 21 | 21
cm
  Week 0 | 7.68 (2.97) | 8.71 (1.57) | 8.24 (1.82) | 8.62 (1.71)
  Week 2 | 8.47 (1.92) | 8.94 (1.51) | 7.63 (2.86) | 7.55 (2.71)

2. Primary Outcome: Injection Duration for the Physiolis Autoinjector at Room Temperature (20° to 27°C) and at Storage Temperature (2° to 8°C) Compared to the Current Autoinjector Ejection Time Specification of Not More Than 10 Seconds
Description: A health care provider administered the injection to the participant, while another recorded the time elapsed during the injection (from the time of autoinjector activation, signaled by the audible "click," until the yellow indicator stopped moving in the autoinjector view window). Injections were administered immediately following removal from the refrigerator (2° to 8°C) or after at least 30 minutes, but no more than 45 minutes, following removal from the refrigerator for the product to reach room temperature (20° to 27°C).
Time Frame: Phase B (Week 4)
Measure: Mean (90% Confidence Interval); unit: seconds
Groups:
- Physiolis Autoinjector 20° to 27°C: Injection performed by health care provider at Week 4 (Visit 3) using Physiolis autoinjector at room temperature (20° to 27°C)
- Physiolis Autoinjector at 2° to 8°C: Injection performed by health care provider at Week 4 (Visit 3) using Physiolis autoinjector at storage temperature (2° to 8°C)
Arm/Group | Physiolis Autoinjector 20° to 27°C | Physiolis Autoinjector at 2° to 8°C
Number analyzed (Participants) | 16 | 18
seconds | 6.66 [6.20 to 7.12] | 6.88 [6.42 to 7.34]

3. Secondary Outcome: Injection Duration for the Current Autoinjector Compared to the Physiolis Autoinjector
Description: as for outcome 2
Time Frame: Phase B (Week 4)
Measure: Mean (90% Confidence Interval); unit: seconds
Groups:
- Current Autoinjector: Injection performed by health care provider at Week 4 (Visit 3) using current autoinjector at storage temperature (2° to 8°C) and room temperature (20° to 27°C)
- Physiolis Autoinjector: Injection performed by health care provider at Week 4 (Visit 3) using Physiolis autoinjector at storage temperature (2° to 8°C) and room temperature (20° to 27°C)
Arm/Group | Current Autoinjector | Physiolis Autoinjector
Number analyzed (Participants) | 47 | 34
seconds | 6.88 [5.85 to 7.90] | 6.78 [6.46 to 7.09]

4. Secondary Outcome: Injection Duration for the Current Autoinjector When Administered at Room Temperature (20° to 27°C) Versus the Storage Temperature (2° to 8°C)
Description: as for outcome 2
Time Frame: Phase B (Week 4)
Measure: Mean (90% Confidence Interval); unit: seconds
Groups:
- Current Autoinjector 20° to 27°C: Injection performed by health care provider at Week 4 (Visit 3) using current autoinjector at room temperature (20° to 27°C)
- Current Autoinjector 2° to 8°C: Injection performed by health care provider at Week 4 (Visit 3) using current autoinjector at storage temperature (2° to 8°C)
Arm/Group | Current Autoinjector 20° to 27°C | Current Autoinjector 2° to 8°C
Number analyzed (Participants) | 20 | 27
seconds | 6.32 [4.35 to 8.29] | 7.29 [6.16 to 8.42]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 70 days following the last treatment. Serious adverse events were collected from the time the participant signed the informed consent.
Description: Those participants that continued on adalimumab therapy after the end of the study were not required to complete the 70-day follow-up.
Groups:
- Current Syringe: Self-injection using current syringe at Week 0 (Visit 1) or Week 2 (Visit 2) (Phase A)
- Physiolis Syringe: Self-injection using Physiolis syringe at Week 0 (Visit 1) or Week 2 (Visit 2) (Phase A)
- Current Autoinjector: Self-injection using current autoinjector at Week 0 (Visit 1) or Week 2 (Visit 2) (Phase A)
- Physiolis Autoinjector: Self-injection using Physiolis autoinjector at Week 0 or Week 2 (Visit 2) (Phase A)
Arm/Group | Current Syringe | Physiolis Syringe | Current Autoinjector | Physiolis Autoinjector | Physiolis Autoinjector at 2° to 8°C | Current Autoinjector 2° to 8°C | Physiolis Autoinjector 20° to 27°C | Current Autoinjector 20° to 27°C
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42 | 0/42 | 0/41 | 0/18 | 0/27 | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 3/40 | 0/42 | 3/42 | 4/41 | 0/18 | 1/27 | 0/16 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Current Syringe (N=40) | Physiolis Syringe (N=42) | Current Autoinjector (N=42) | Physiolis Autoinjector (N=41) | Physiolis Autoinjector at 2° to 8°C (N=18) | Current Autoinjector 2° to 8°C (N=27) | Physiolis Autoinjector 20° to 27°C (N=16) | Current Autoinjector 20° to 27°C (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Odema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.